CLINICAL TRIAL: NCT06388850
Title: Evaluation of the School-based Healthy Relationships Project for Primary Prevention of Child Sexual Abuse Among Children Pre-K Through 5th Grade
Brief Title: Evaluation of HRP Among Pre-K Through 5th Grade
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Responsible Party: Principal Investigator, Beth Molnar, Professor, Northeastern University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5U01CE003393-03 (NIH)
Record Dates: First submitted 2024-03-20; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Child Sexual Abuse

STUDY DESIGN:
Intervention Model Description: A stepped wedge cluster randomized clinical trial design will be used to assess the efficacy of two linked curricula of the Healthy Relationships Project (HRP): Care for Kids (Pre-K through 2nd Grade) and We Care Elementary (3rd through 5th Grade). The HRP includes a 1.5 hour training for school staff prior to implementation, six 30-minute classroom lessons delivered to students once per week for 6 weeks, and 3 caregiver workshops.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Schools receiving HRP programming in pre-k through 5th-grade classrooms.
  Interventions: Behavioral: Healthy Relationships Project
- Control Group (No Intervention): Schools that have not received HRP programming. Schools in the control group will continue their normal standard of care for CSA prevention.

INTERVENTIONS:
Behavioral: Healthy Relationships Project — The Healthy Relationships Project (HRP), created by the community-based organization Prevent Child Abuse Vermont (PCAVT), will be the focus of this rigorous evaluation study. The program is fully manualized with a widely accepted curriculum designed for Pre-K to 2nd graders (Care for Kids) and 3rd to 6th graders (We Care Elementary, though implementation will stop at 5th grade for this study). The HRP uses an upstream universal public health approach for the primary prevention of child and youth perpetration of child sexual abuse with developmentally appropriate intervention elements for children, faculty and staff at their schools, and for their caregivers.
  Arms: Intervention Group

SUMMARY:
This study is a rigorous experimental evaluation of an existing manualized universal child sexual abuse primary prevention program with a history of 30+ years of implementation across 30 states and robust pilot data.

DETAILED DESCRIPTION:
The Healthy Relationships Project (HRP) created, modified and run by the organization Prevent Child Abuse Vermont, has been delivering CSA primary prevention curricula since 1990 with implementation across 30 U.S. States, including statewide in Vermont. During those decades, substantiated cases per year in Vermont dropped 61%, and the number of child perpetrators per year dropped 69%. Addressing Research Priority 1, implementation of the HRP in Pre-K through 5th grade will be rigorously evaluated in a mixed-methods stepped wedge randomized trial design with 16 public charter schools in three high-need wards in Washington, DC. The School Safety Omnibus Amendment Act of 2018 was enacted to obligate DC schools to prevent and address student sexual abuse. The partner organization, Safe Shores, the Child Advocacy Center (CAC) for DC, has implemented HRP in public charter schools with success; the opportunity remains to conduct this trial in schools where it has not been delivered and increase its feasibility via established trust with the district and schools. The findings about its efficacy will potentially place the HRP into the echelon of evidence-based programs that many schools seek to use, especially those mandated to deliver CSA prevention programming. Data from Safe Shores, the CAC that receives reports of suspected child abuse from all Washington, DC public schools, will be utilized as the primary outcome, including the numbers and types of CSA investigations and other services provided by the CAC involving the participating schools, which include forensic services, family advocacy, case management and more. More commonly utilized measures of improvements in protective behaviors, self-efficacy, knowledge and disclosure will be collected from caregivers and teachers. Qualitative research will be included to assess the strengths and weaknesses of intervention rollout, fidelity monitoring, lessons learned and sustainability. This innovative and novel mixed methods evaluation study will move the science of child sexual abuse prevention research forward with a community-based participatory research partnership between scientists in family violence prevention research, professionals at community-based organizations, and participating public elementary schools in high-need urban areas. In summary, a rigorous experimental evaluation of an existing universal primary prevention program with a history of 30+ years of implementation across 30 states and robust pilot data will be conducted.

Specific Aims:

Aim 1: Test the efficacy of the Healthy Relationships Program in reducing reports of child sexual abuse by implementing a stepped wedge randomized trial design. Sixteen (minimum, possibly up to 24) public schools/public charter schools in Washington D.C. serving approximately 8,960 (or 13,440 with 24 schools) urban, ethnically diverse children in grades Pre-K through 5 will transition from waitlist to active intervention condition in 6-month intervals using stratified randomization. It is hypothesized that over 1 year, rates of CSA reports from schools receiving the HRP may be lower relative to reports from schools that did not receive the HRP or may be higher given increased awareness provided by the program. These reports will be generated by data collected by Safe Shores, the Child Advocacy Center (CAC), whose multidisciplinary teams support Washington, DC's children who have been the subject of a child abuse report, as well as their families.

Aim 2: Test the efficacy of the HRP in reducing theory-based intervention mechanisms among caregivers and teachers. The investigators expect over 1 year, caregivers of children receiving the HRP and teachers/facilitators will have improved knowledge of CSA, knowledge of grooming behaviors, parental monitoring, internet safety, parent-child communication about consent, and self-efficacy for CSA protection, relative to baseline. The investigators expect over 1 year, teachers and social workers implementing the HRP curriculum, as well as caregivers of the children receiving it, will have improved CSA knowledge, self-efficacy for reporting, comfort with CSA education and prevention of CSA behaviors by children, relative to baseline. The investigators plan to measure these mechanisms via online surveys distributed to all teachers and caregivers of children in grades Pre-K through 5. The surveys will be distributed a total of 5 times to meet the requirements of the stepped wedge randomized trial design.

Aim 3: Conduct a qualitative evaluation of the sustainability of the HRP, with ongoing input from community stakeholders. The investigators will interview school and community-based stakeholders to understand the perceived capacity, buy-in, and impact of ongoing implementation of the HRP program through school-community partnerships. The investigators hypothesize that important sustainability characteristics can be identified to facilitate future dissemination efforts. These interviews will happen both before and after the implementation of the HRP at the participating schools.

ELIGIBILITY:
Inclusion Criteria:

* Public schools/public charter schools in high-need wards of Washington D.C.
* Enrolling children in pre-k through 5th grade

Exclusion Criteria:

* Private schools
* School in non high-need wards

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Reports of child sexual abuse | Every month, over 2 years
  The number and proportion of child sexual abuse reports per school, per grade, to a Child Advocacy Center (CAC) in Washington, DC will be shared with the investigators bi-monthly and will serve as the primary outcome to test the efficacy of the HRP in prevention of incidence of CSA.

SECONDARY OUTCOMES:
The Parental Knowledge Scale (PKS) | Every 6 months, over 2 years
  This measure measures caregiver monitoring behaviors. Parental knowledge is measured on a 5-point Likert scale, with 1=strongly disagree; 2=disagree; 3=neither agree nor disagree; 4=agree; 5=strongly agree 9=Don't know/Prefer not to answer. Participants are asked to respond to a list of eight statements. A score is determined by the sum of answers for all eight statements, with higher scores indicating higher monitoring behavior.
The Parental Discussions about Sex Abuse Scale (PDSAS) | Every 6 months, over 2 years
  This scale is used to assess caregiver-child communication about consent and CSA topics. This scale uses 16 statements asking participants to indicate their level and comfort discussing CSA topics with their children. Participants are asked to respond to the question: "Have you spoken to your child about this topic and what degree of comfort did you feel?" with answer choices 1=Never, 2=Yes, but I felt uncomfortable with the discussion, 3=Yes, and I felt at ease with the discussion, and 9=Don't know/Prefer not to answer. A score is determined by the sum of answers for all statements, with higher scores indicating higher comfort and engagement with discussions about sexual abuse.
The adapted Parenting Self Agency (PSAM) | Every 6 months, over 2 years
  This scale is used to assess caregiver self-efficacy for protecting their child from CSA. Participants are asked to respond to six statements with a 5-point Likert scale where 1=strongly disagree; 2=disagree; 3=neither agree nor disagree; 4=agree; 5=strongly agree 9=Don't know/Prefer not to answer. This scale is scored as a sum of answers across all statements. A higher score indicates a higher self-efficacy.
The Parent Knowledge Questionnaire (PKQ) | Every 6 months, over 2 years
  This scale assesses how a caregiver imagines their child would respond to various instances of CSA-related behaviors. Participants are asked to respond to the question: "WITHOUT ASKING YOUR CHILD; how do you think your child would answer the following questions?" There are nine statements with answer choices for 1=True; 2=False; 3=Don't know; 4=Prefer not to answer. The scale is scored by summing the number of "1" responses selected. A higher count of "1" responses indicates a higher CSA knowledge.
HRP evaluation | Every 6 months, over 2 years
  Items from the previously implemented post-intervention survey from the HRP evaluation (HRPS) will be administered to assess knowledge of CSA grooming behaviors and internet safety. Participants are asked to state the agreement/disagreement with 18 statements with answer choices for 1=strongly disagree; 2=disagree; 3=neither agree nor disagree; 4=agree; 5=strongly agree 9=Don't know/Prefer not to answer.
The CSA Myths Scale | Every 6 months, over 2 years
  This scale measures the acceptance of common CSA myths. School staff participating in the study will be asked to state their level of agreement with 25 statements with answer choices for 1=strongly disagree; 2=disagree; 3=neither agree nor disagree; 4=agree; 5=strongly agree 9=Don't know/Prefer not to answer. A score is determined by a sum of the statements, with a higher score indicating higher endorsement of CSA myths.
The Teachers' Reporting Attitudes Scale for Child Sexual Abuse (TRAS-CSA) | Every 6 months, over 2 years
  This scale tests three constructs: commitment, concerns, and confidence related to reporting behaviors which are independently and equally important in the evaluation of teacher preparation and training. School staff participating in the study will be asked to state their level of agreement with 20 statements with answer choices for 1=strongly disagree; 2=disagree; 3=neither agree nor disagree; 4=agree; 5=strongly agree 9=Don't know/Prefer not to answer. A score is determined by a sum of the answers for all statements, with a higher score indicating more positive CSA reporting behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- Safe Shores, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No